CLINICAL TRIAL: NCT03875196
Title: The Effect Of Pelvic Floor Muscle Training With Bıofeedback And Extracorporeal Magnetic Innervation On The Urinary Symptoms, Sexual Function And Quality Of Life Of Women With Stress Urinary Incontinence
Brief Title: The Effect Of Pelvic Floor Muscle Training With Biofeedback And Extracorporeal Magnetic Innervation On The Urinary Symptoms, Sexual Function And Quality Of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, sureyya gumussoy, associate professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-7/5
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Urinary Incontinence
Keywords: Stress urinary incontinence; quality of life; sexual function
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Masking Description: The sample of the research is comprised of patients diagnosed with stress urinary incontinence and volunteered for participating in the study with the following specifications: with pelvic floor power 2 and over, sexually active and no restrictions for the magnetic chair treatment. Patients with the following conditions were excluded: prosthesis, other implanted metallic devices, cardiac pacemaker, arrhythmia, pelvic malignancies, under radiotherapy, pelvic floor defect, previous surgery for urinary incontinence, neurological diseases and pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biyofeedback (Experimental): the patients underwent 16 sessions of biofeedback-assisted pelvic floor muscle training over 8 weeks for 20 minutes
  Interventions: Device: Pelvic Floor Muscle Training With Biofeedback
- Extracorporeal Magnetic Innervation (Experimental): the patients underwent 16 sessions of biofeedback-assisted pelvic floor muscle training over 8 weeks for 20 minutes and the Extracorporeal Magnetic Innervation application was made for 20 minutes
  Interventions: Device: Pelvic Floor Muscle Training With Biofeedback; Device: Extracorporeal Magnetic Innervation

INTERVENTIONS:
Device: Pelvic Floor Muscle Training With Biofeedback — Biyofeedback: The Biyofeedback allows the patient to see the results of her behavior immediately By a perineometer device or electromyelography that is placed in the vagina, the patient sees how she hears the pelvic floor muscles, hears the sound or hears her voice, and detects how much she needs to contract.
Device: Extracorporeal Magnetic Innervation — Extracorporeal Magnetic Innervation: The patients are seated in a special chair connected to an external power unit and a magnetic field generator inside with their clothes on. In order to coincide the spreading magnetic field with pelvic floor muscles, the urethral and anal sphincters, the perineum of the patients should be placed in the center of the chair. In this way, the perineum tissues are stimulated by emitted magnetic field waves. Thus no electrical current passes through the device to the patient's body and the patient is exposed to only the magnetic current.
  Arms: Extracorporeal Magnetic Innervation

SUMMARY:
The effect of Pelvic Floor Muscle Training with Biofeedback and Extracorporeal Magnetic Innervation on the Urinary Symptoms, Sexual Function and Quality of Life of Women with Stress Urinary Incontinence

DETAILED DESCRIPTION:
Introduction and hypothesis: This research was made in order to analyze the impact of the with with Electromyelographic-Biyofeedback added Extracorporeal Magnetic Innervation technique performed on the urinary symptoms, quality of life and sexual function of women with stress urinary incontinence.

Methods: The research type is a pre-test and post-test randomized controlled with experimental nature. The research sample consists of 26 patients in the Biyofeedback group and 25 patients in the with Electromyelographic-Biyofeedback added Extracorporeal Magnetic Innervation group who were examined in the urogynecology policlinics and diagnosed with stress urinary incontinence. between September 2015 and September 2016. At the first meeting, the case report form is filled and the following list is applied for each patience: incontinence life quality scale, female sexual function scale, Q-type test, residue urine volume, one-hour pad test, perineometer, muscle force measurement with Modified Oxford Scale and a three-day bladder diary. Moreover, the Electromyelographic-Biyofeedback was applied to the first group in the clinic for 20 minutes two days a week for eight weeks. The Electromyelographic-Biyofeedback following with 20 minutes Extracorporeal Magnetic Innervation was applied to the second group in the clinic for 20 minutes two days a week for eight weeks. The list applied at the first meeting were repeated after eight weeks.

ELIGIBILITY:
Inclusion Criteria

* patients diagnosed with stress urinary incontinence
* with pelvic floor power 2 and over,
* sexually active and no restrictions for the magnetic chair treatment.

Exclusion Criteria:

patients with

* prosthesis,
* other implanted metallic devices,
* cardiac pacemaker,
* arrhythmia,
* pelvic malignancies,
* under radiotherapy,
* pelvic floor defect,
* previous surgery for urinary incontinence,
* neurological diseases
* pregnancy.

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Strength with Perineometer | In the first encounter and After eight weeks
  Perineometer: It is a vaginal dynamometer used for objective evaluation of pelvic floor muscle strength during its contractions. The intravaginal pressure unit is, cmH2O İn. The pelvic floor muscle strength is evaluated by placing the vaginal probe 3 cm deep inside vagina. The nominal measurement range is 30-60 cmH2O. Pressure may decrease to 0-5 cmH2O in patients with weak pelvic floor muscles
Pelvic Floor Muscle Strength with Modified Oxford Scale | In the first encounter and After eight weeks
  Modified Oxford Scale:
  Grade 0: No contraction. Grade 1: Contraction is minimal. The patient can hold the fingers under 1 second.
  Grade 2: Contraction is poor. There is no elevation in the fingers. The patient can hold the fingers for 1-3 seconds.
  Grade 3: The fingers of the therapist are elevated to the posterior vaginal wall with contraction. There is a minimal pressure and the patient can hold the fingers for 4-6 seconds.
  Grade 4: The fingers of the therapist are elevated to the posterior vaginal wall. There is a sense of intensive pressure on the fingers. The patient can hold the fingers for 7-9 seconds.
  Grade 5: A strong contraction lasting for 9 seconds and a great resistance against the fingers of the therapist.
Incontinence Quality of Life | In the first encounter and After eight weeks
  The quality of life of the patients was measured by the Incontinence Quality of Life Questionnaire IQOL consists of 22 questions and three subscales: behavior limitations (1st, 2nd, 3rd, 4th, 10th, 11th, 13th, 20th items), the psychosocial influence (5th, 6th, 7th, 9th, 15th, 16th, 17th, 21st, 22nd items) and the social isolation (8th, 12th, 14th, 18th, 19th items). All items in I-QOL are evaluated with a five-category Likert-type scale: 1= very much, 2= quite, 3= moderate, 4= somewhat, 5= not at all. The calculated total score is converted to a value between 0 to 100 to interpret the results easily. The increased score obtained from the scale indicates an increase in quality of life.
Sexual Function | In the first encounter and After eight weeks
  Female Sexual Function Index consists of 19 items and 6 subscales developed by Rosen et al. in 2000 to assess female sexual function in the USA. In this scale, sexual problems or functions in the last four weeks are assessed. Of the items in the scale, 3-14 and 15-19 are rated on a 6-point Likert scale ranging between 0 and 5, and the rest are rated on a 5-point Likert scale ranging between 1 and 5. The scoring of the scale items is different. While the items 1, 2, 15 and 16 are rated as 5-4-3-2-1, the other items are scored as 0-1-2-3-4-5. The total score for the overall scale is calculated by multiplying the scores obtained from the subscales by the factor loads. The lowest and highest achievable scores from the scale are 2.0 and 36.0 respectively.
The amount of leakage | In the first encounter and After eight weeks
  Pad Test: In the study, a one-hour pad test standardized by the International Continence Society was applied to the patients and it was evaluated as the following:
  <2 gr- Dry 2-10 gr- Mild/Moderate Urinary Incontinence 10-50 gr- Severe Urinary Incontinence > 50 gr- Very Severe Urinary Incontinence

CONTACTS AND LOCATIONS:
Overall Officials: oya kavlak, proffesor, Study Director — Ege University; ahmet özgür yeniel, assosiate prf, Study Chair — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No